CLINICAL TRIAL: NCT04882137
Title: A Study to Understand the Barriers in Referring Adolescent Women for the Etonogestrel Implant and to Evaluate Whether Intensive Coaching on the Management of Common Side Effects of the Implant Influences Referrals for the Implant.
Brief Title: Barriers to Referring Adolescent Women for Etonogestrel Implant.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was stopped due to shifted research priorities by funder
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lonna Gordon, Chief, Adolescent Medicine, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1692814
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Education (No Intervention): Pediatric Providers in this arm will receive a continuing medical education on etonogestrel contractive implant but will not receive specialist coaching on how to manage side effects.
- Standard Education plus Coaching (Experimental): Pediatric Providers in this arm will receive a continuing medical education program on etonogestrel contraceptive implant. Providers in this arm will also receive a tip-sheet on how to manage side effects as well as a number to directly access a specialist who places them if needed.
  Interventions: Behavioral: Education plus Coaching

INTERVENTIONS:
Behavioral: Education plus Coaching — Providers in Intervention group will receive standard education (1.5 hr CME), a tip sheet on how to manage side effects for quick reference and a number to directly reach a provider experienced with managing etonogestrel side effects with questions regarding how to manage side effects.
  Arms: Standard Education plus Coaching

SUMMARY:
This study seeks to understand how much pediatric providers in Central Florida know about the etonogestrel contraceptive implant. The investigators also seek to understand the barriers that may prevent them from referring adolescent women for this highly effective and recommended method of contraception. Finally the study will consider if an expanded education and coaching improves their ability to referring patients for this method of birth control.

DETAILED DESCRIPTION:
This study is comprised of two phases. During the first phase 500 medical providers who provide care to adolescents will be recruited to complete a 30 question anonymous survey that evaluates their attitudes towards recommending and referring for adolescent women for the etonogestrel contraceptive device. This survey will also test participant's knowledge of indications, side effects and side effect management related to this contraceptive device as well.

During phase 2, 100 pediatric providers will be randomized to two groups. One group will receive standard continuing medical education on the use of the etonogestrel device in adolescents focusing on themes that emerged as knowledge deficits in phase 1. The other group will receive standard continuing medical education plus continued coaching on management of medication side effects. The referring patterns of physicians in each group will be studied.

ELIGIBILITY:
Inclusion Criteria:

* A primary care provider that cares for children under the age of 18. This includes physician's assistants, advanced nurse practitioners, residents or fellows, and physicians in pediatrics, internal medicine, and family medicine.
* Must currently be practicing in Central Florida.
* Be able to speak and write in English
* For phase two of the study an additional requirement is that you must have a medical license to practice independently in the state of Florida.

Exclusion Criteria:

* Not a primary care provider who cares for children.
* A pediatric provider who only provides specialty care
* Not able to speak or write in English
* For phase two of study does not have a medical license to practice independenly in the State of Florida.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Types of barriers to referral for etonogestrel implant based on questionnaire | 6 months
  Barriers to recommending and referring adolescent women for etonogestrel contraceptive implant
Number of adolescent women referred | 18 months
  Number of adolescent women who were referred for etonogestrel contraceptive implant

SECONDARY OUTCOMES:
Categories of knowledge deficit in pediatric providers based on questionaire | 6 months
  Understanding whether pediatric providers main knowledge deficit around etonogestrel implant is indications, side effects, or decreasing side effects.
Aspects in Coaching that changed pediatric providers' behaviors | 18 months
  Qualitative analysis on which parts of coaching or standard intervention were most considered in referring.

CONTACTS AND LOCATIONS:
Overall Officials: Lonna P Gordon, MD, Principal Investigator — Nemours Children's Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT04882137/Prot_000.pdf